CLINICAL TRIAL: NCT05075330
Title: SMART Trial: Reducing Stigma Towards Opioid Use Disorder at the Community Level
Brief Title: SMART Trial: Community Stigma Reduction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Karen Derefinko, PhD (Other)
Collaborators: National Center for Complementary and Integrative Health (NCCIH) (NIH)
Responsible Party: Sponsor-Investigator, Karen Derefinko, PhD, Associate Professor, University of Tennessee
Organization: University of Tennessee (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 21-08181-XP
Record Dates: First submitted 2021-09-14; First posted 2021-10-12 (Actual); Last update posted 2022-03-18 (Actual); Status verified 2022-03

CONDITIONS: Opioid-use Disorder; Stigma, Social
Keywords: stigma; opioid use disorder; community
MeSH Terms: conditions — Opioid-Related Disorders; Social Stigma

STUDY DESIGN:
Intervention Model Description: Participants assigned to intervention or control based on zip code of primary residence.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Participants who live in the Orange Mound community of Memphis. Billboards targeting stigma reduction were posted in the community for one month.
  Interventions: Behavioral: Opioid Use Disorder Stigma Reduction
- Control (No Intervention): Participants who live in the Frayser community of Memphis. No billboards (intervention) were placed here.

INTERVENTIONS:
Behavioral: Opioid Use Disorder Stigma Reduction — Billboards with destigmatizing language regarding opioid use disorder placed in the community.
  Arms: Intervention

SUMMARY:
The goal of this project is to engage community members from two low-income African American communities (N=200) in a survey study that assesses stigma toward those with Opioid Use Disorder (OUD). Those from the intervention community will be subject to a stigma reduction campaign via billboards. Those from the control community will not. Stigma will be re-assessed following the period of the campaign.

ELIGIBILITY:
Inclusion Criteria:

* Identify as African American or Mixed race
* Reside in Frayser or Orange Mound Communities
* Access to telephone for follow-up assessment

Exclusion Criteria:

* Unable to understand consent procedures

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 199 (Actual)
Dates: Start 2021-06-16 (Actual); Primary Completion 2021-08-19 (Actual); Study Completion 2021-08-19 (Actual)

PRIMARY OUTCOMES:
Stigma score | Change from baseline stigma score at 8 weeks
  Pre- and post-intervention stigma assessments using the Exposure to Drug Users Index, Drug Use Stigmatization Scale, and the Stigma of Drug Users Scale

CONTACTS AND LOCATIONS:
Overall Officials: Karen Derefinko, PhD, Principal Investigator — University of Tennessee
Locations (1):
- University of Tennessee Health Science Center, Memphis, Tennessee, United States

IPD SHARING:
Plan to Share IPD: Yes
Time Frame: Available by end of 2021.